CLINICAL TRIAL: NCT02676869
Title: A Multicentre, Open Label, Dose Escalation, Phase 1 Study in Patients With Unresectable or Metastatic Melanoma Receiving IMP321 (LAG-3Ig Fusion Protein-eftilagimod Alpha) as an Adjunctive Therapy to Anti-PD-1 Therapy With Pembrolizumab
Brief Title: Phase 1 Study of IMP321 (Eftilagimod Alpha) Adjuvant to Anti-PD-1 Therapy in Unresectable or Metastatic Melanoma
Acronym: TACTI-mel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immutep Australia Pty. Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMP321-P012
Record Dates: First submitted 2016-02-02; First posted 2016-02-08 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Stage IV Melanoma; Stage III Melanoma
MeSH Terms: conditions — Melanoma | interventions — soluble LAG-3 protein, human; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Study is an open label, dose finding study consisting of 2 parts. In part A, the dose is escalated following the protocol-defined safety observation period of the previous cohort. Patients will receive 9 cycles Pembrolizumab in combination with IMP321. In part B, the dose was defined based on the dose escalation. The treatment duration will be expanded to 19 cycles in the combined treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMP321 dose escalation (Experimental): IMP321 administered fortnightly in addition to SOC pembrolizumab.
  Interventions: Drug: IMP321 (eftilagimod alpha); Drug: Pembrolizumab

INTERVENTIONS:
Drug: IMP321 (eftilagimod alpha) — Part A: Single subcutaneous injections of 1 mg (cohort 1), 6 mg (cohort 2) or 30 mg (cohort 3) of IMP321 administered every 2 weeks
  Part B: Single subcutaneous injections of 30 mg of IMP321 administered every 2 weeks
  Other Names: Eftilagimod alpha
Drug: Pembrolizumab — Administered according to the approved label.

SUMMARY:
The purpose of this study is to determine the safety, tolerability and recommended phase 2 dose of a new drug, known as IMP321, in combination with pembrolizumab when given to patients with unresectable or metastatic melanoma.

ELIGIBILITY:
Main Inclusion Criteria

* Histologically confirmed diagnosis of locally advanced (unresectable Stage III) or metastatic (Stage IV) melanoma
* Currently receiving anti-PD-1 therapy with pembrolizumab and after 3 cycles achieved asymptomatic irPD (slowly progressive, not requiring urgent intervention, and stable performance status) or sub-optimal response (irSD, irPR) as demonstrated in imaging assessments performed within 6 weeks prior to study start
* Female or male 18 years of age or above
* ECOG performance status 0-1
* Evidence of measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 10. Adequate Laboratory criteria

Main Exclusion Criteria

* More than four prior lines of therapies for advanced or metastatic disease.
* Prior PD-1/PDL-1 targeted therapy
* Currently receiving treatment with another investigational drug, or less than 4 weeks since ending treatment on another investigational drug
* Currently receiving systemic chemotherapy, targeted small molecule therapy, radiotherapy, or biological cancer therapy (other than pembrolizumab) or less than 4 weeks since completion of these therapies and first dose of study treatment
* History of irAEs from ipilimumab of CTCAE Grade 4 requiring steroid treatment
* Known cerebral or leptomeningeal metastases
* Serious intercurrent infection within 4 weeks prior to first dose of study treatment
* Active acute or chronic infection
* History or evidence of interstitial lung disease or active non-infectious pneumonitis
* Active auto-immune disease requiring immunosuppressive therapy
* HIV positivity, active hepatitis B or hepatitis C
* Continuous systemic treatment with either corticosteroids or other immunosuppressive medications within 4 weeks prior to first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To assess the recommended phase 2 dose | From the time of inform consent form signature until 30 days after end of treatment
To asses frequency of adverse events | From the time of inform consent form signature until 30 days after end of treatment
To asses severity of adverse events | From the time of inform consent form signature until 30 days after end of treatment
To asses duration of adverse events | From the time of inform consent form signature until 30 days after end of treatment

SECONDARY OUTCOMES:
Best overall response rate (ORR) to irRC and RECIST 1.1 | From the time of inform consent form signature until 30 days after end of treatment.
Time to next treatment (TTNT) | Up to 12 months
Progression-free survival | Up to 12 months
Overall survival (part B only) | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Royal Brisbane Womens Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Greenslopes Private Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Ballarat Hospital, Ballarat, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided